CLINICAL TRIAL: NCT01528995
Title: A Blinded Randomized Controlled Clinical Trial Comparing Sacral Nerve Modulation and Anal Bulking Injections as Treatment for Fecal Incontinence After Obstetric Anal Sphincter Injuries (OASIS).
Brief Title: Treatment of Fecal Incontinence After Obstetric Anal Sphincter Injuries
Acronym: KISS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011/|1300/REKnord
Record Dates: First submitted 2012-01-26; First posted 2012-02-08 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Fecal Incontinence
Keywords: fecal incontinence; anal incontinence; obstetric sphincter injuries; OASIS; double incontinence; urinary incontinence; sexual function; sacral nerve modulation; sacral nerve stimulation; Interstim; anal bulking injections; Permacol
MeSH Terms: conditions — Fecal Incontinence; Encopresis; Urinary Incontinence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- sacral nerve modulation (Active Comparator): Implantation of Interstim II-3058 impulse generator after positive PNE test. Randomized controlled trial.
  Interventions: Device: Medtronic Interstim II-3058
- anal bulking agents (Active Comparator): anal injection with Permacol after positive PNE test. Randomized controlled trial.
  Interventions: Procedure: Anal bulking injection
- Anal bulking agents (Active Comparator): Anal injection with Permacol after negative PNE test. cohort study.
  Interventions: Procedure: Anal bulking injection

INTERVENTIONS:
Device: Medtronic Interstim II-3058 — impulse generator
  Arms: sacral nerve modulation
Procedure: Anal bulking injection — Permacol injection:
  four submucosal injections are administered at the 12, 3, 6 and 9 o'clock positions, above the level of the dentate line. The injection produces a bulge in the mucosa
  Arms: Anal bulking agents; anal bulking agents

SUMMARY:
Fecal incontinence (FI), the involuntary loss of solid or liquid stool, is a stigmatising condition. It can have a distressing impact and restriction on quality of life. Obstetric-related fecal incontinence may occur early after childbirth. Previous obstetric injury is a major cause of fecal incontinence in older women.

When conservative treatment fails, surgery may be an option. Both sacral nerve modulation and anal bulking injections is minimal invasive surgical alternatives. Step one in SNM is a trial period of temporary stimulation. If the test is successful, the patient can have an implantable stimulator (step 2). Transanal submucosal bulking injection of collagen is also a possible treatment option and can be an effective treatment for faecal incontinence.

The purpose of this study is to compare the efficacy of sacral nerve stimulation to anal bulking injections in women with fecal incontinence after obstetric sphincter injuries (OASIS), through a multicenter blinded, randomized controlled trial.

DETAILED DESCRIPTION:
Obstetric anal sphincter injuries (OASIS) is the most common cause of fecal incontinence (FI) in women. Obstetric-related FI may occur early after childbirth. Previous obstetric injury is also a major cause of FI in older women, and risk of FI increases with time and further childbirths. FI is involuntary loss of solid or liquid stool. Symptoms range from fecal urgency, soiling, to daily passive or urge fecal incontinence. FI is a stigmatizing condition. It can have a distressing impact and restriction on quality of life, including isolation and depression.

Tears during delivery is classified (Sultan) as first degree tears including vaginal epithelium, second degree tears into the perineal muscle, third degree involving the anal sphincter complex and fourth degree including sphincter complex and anorectal epithelium. OASIS includes third and fourth degrees tears.

First line of therapy of FI is conservative treatment including drug therapy and "biofeedback". If conservative treatment fails, surgery may be an option. Traditionally elective secondary sphincter repair has been performed at least once. Sphincter repair may improve symptoms in short time, but efficacy deteriorates with time.

Other minimal invasive surgical alternatives includes sacral nerve modulation (SNM) and anal bulking injection. Sacral nerve modulation involves stimulating the sacral nerves, usually S3 or S4. Step one is a trial period of temporary stimulation (PNE test). If the test is successful, the patient can have an implantable stimulator (step 2) to modulate sacral nerve function. SNM is also beneficial for treating FI after OASIS, and SNM is a alternative to secondary sphincter repair. SNM should possibly be preferred second line treatment also after sphincter tears related FI. Transanal submucosal bulking injection of collagen is also a possible treatment option and can be an effective treatment for both anal and fecal incontinence.

The purpose of this study is to compare the efficacy of sacral nerve modulation to anal bulking injections in women with fecal incontinence after OASIS through a Scandinavian multicenter single-blinded, randomized controlled trial.

To answer the research question, we will include 66-86 women with FI after OASIS. Sphincter defects are classified using three dimensional endoanal ultrasonography. Pelvic floor function including FI is registered using validated questionnaires. All women eligible for inclusion is PNE-tested for three weeks. The purpose of this cohort analysis, is to examine the possible effect of SNM in women with sphincter defects, and the hypothesis is that there is no relation between sphincter defect classified using tree dimensional ultrasound and efficacy of SNM.

Women with more than 50 % symptom reduction during PNE test (positive PNE test), is further randomized and allocated 1:1 into one of two arms with 28 participants. One group is allocated to implantation of permanent impulse generator, Interstim II-3058 and the other group is allocated to anal sub mucosal bulking injection of collagen, Permacol. The purpose of this study is to compare the efficacy of SNM to anal bulking injection. The hypothesis is that SNM provides a mean change in improvement in St Marks Incontinence score of more than 4 compared to the anal bulking group. This study is designed as a multicenter single-blinded, randomized controlled trial.

Women with less than 50 % symptom reduction (15-28, negative PNE test), is treated in a third arm with anal bulking injection. The purpose of this cohort study, is to examine the efficacy of anal bulking injection in women suffering from FI after sphincter tears, excluded from further treatment with SNM.

ELIGIBILITY:
Inclusion Criteria:

* fecal incontinence after OASIS
* St Marks score > 8
* failure of conservative treatment

Exclusion Criteria:

* pregnancy
* immunosuppressed
* former major pelvic surgery or irradiation
* Rectal prolapse
* complex fistula
* IBD
* Lateral sphincterotomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2012-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
change in St Marks incontinence score | 6 month after treatment
  Vaizey Incontinence Score A scale from 0-24 where 0 = perfect continence and 24 = complete incontinence. 3, 6 and 12 months

SECONDARY OUTCOMES:
change in number of fecal incontinence and urgency episodes per week | 3 and 6 month after treatment
change in Quality of life assessment (Rockwood- Fecal incontinence quality of life ) | 3 and 6 month
  change in FIQL and EQ-5D
change in urinary incontinence score (ICIQ-UI SF) | 3 and 6 month
  International consultation on incontinence modular questionnaire, ICIQ-UI Short form, A scale from 0-21 where 0 = perfect continence and 20 = complete incontinence.
change in sexual function | 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stig Norderval, PHD MD, Principal Investigator — University Hospital of North Norway
Locations (1):
- Dep. of Colorectal Surgery, University Hospital of North Norway, Tromsø, Troms, Norway